CLINICAL TRIAL: NCT05147584
Title: Trans-abdominal Fetal Pulse Oximetry: PILOT 1
Brief Title: Trans-abdominal Fetal Pulse Oximetry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device Modifications and Relocation of Principal Investigator
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PILOT 1
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Fetal Hypoxia; Fetal Distress; Fetal Acidemia; Fetal or Neonatal Effect of Complication of Labor
MeSH Terms: conditions — Fetal Hypoxia; Fetal Distress

STUDY DESIGN:
Intervention Model Description: This is a prospective, investigator-blinded study that is for data collection only. The primary purpose is to verify accuracy during the training of the algorithm by comparing the external sensor to a known internal sensor.
Masking Description: Results of either the external sensor or the internal sensor will not be shown to the subject, the care provider, or the investigator and will not be used to guide or alter patient management. The "outcomes assessor" will review the subject CTG and sensor data retrospectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Interventional/Observational (Experimental): The internal and external oxygen sensors will be used to record fetal oxygen during active labor and these will be be compared to the CTG retrospectively.
  Interventions: Device: Dual fetal oxygen sensors

INTERVENTIONS:
Device: Dual fetal oxygen sensors — Placement of both internal and external fetal oxygen sensors

SUMMARY:
The Raydiant Oximetry Sensing System (Lumerah) is a non-invasive fetal pulse oximeter that measures fetal arterial oxygen saturation using safe, non-invasive, transabdominal near-infrared spectroscopy. Lumerah is intended as an adjunct to cardiotocography by detecting decreases in fetal oxygenation.

DETAILED DESCRIPTION:
Raydiant Oximetry, Inc. is developing a novel and non-invasive fetal pulse oximetry device to fundamentally improve how fetuses are monitored during labor. The Raydiant Oximetry Sensing System (Lumerah) is a fetal pulse oximeter that measures fetal arterial oxygen saturation using safe, non-invasive, transabdominal near-infrared spectroscopy. Lumerah performs its measurements without the requirement for transvaginal placement and its associated risks. Lumerah is intended as an adjunct to cardiotocography by detecting fetal oxygen deprivation which is both life-threatening to the fetus and can lead to the irreversibly debilitating consequences of newborn metabolic acidosis. The severe consequences associated with newborn metabolic acidosis and the lack of availability of an effective tool to support its early diagnosis led to the development of Lumerah.

In this study, women in labor will be simultaneously monitored with proven (previously FDA-approved) technology as a "ground truth". These women will be simultaneously monitored with both an external and internal oxygen sensor. Obstetric health-care providers are blinded to oximetry data presented by both devices; therefore, clinical decisions regarding interventions are made based on the standard factors, including cardiotocography. The primary efficacy analysis will be performed retrospectively by comparing data of fetal oxygenation displayed and recorded by both devices. Results of either the Lumerah external sensor or the internal sensor will not be used to guide or alter patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable to provide informed consent
2. Age > 18 years
3. BMI < 50 (with no more than 4 cm between maternal skin and fetal skin)
4. Gestational age > 36 weeks
5. Singleton pregnancy
6. Vertex presentation
7. Active labor
8. Category I or Category II tracings
9. Ruptured amniotic sac with cervical dilation of >2 cm and a station of -2 or lower

Exclusion Criteria:

1. Age <18 years
2. BMI > 50 third trimester
3. Gestational age < 36 weeks
4. Multiple gestation
5. Nonvertex fetal presentation
6. Suspected vasa previa
7. Latent labor
8. Category III CTG tracing (i.e., need for immediate delivery)
9. Fetal anomalies and/or chromosomal disorders
10. Chorioamnionitis
11. Placenta Previa
12. History of HIV, Genital Herpes, or other infection precluding internal monitoring
13. Unable to provide informed consent (e.g., cognitively impaired)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are in labor
Enrollment: 31 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosen, MD, Study Director — Raydiant Oximetry
Locations (1):
- University of Texas Medical Branch (UTMB), Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is for device development only, there is no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional/Observational
Started | 31
Completed | 23
Not Completed | 8
Not completed — Subjects consented but did not fully meet inclusion /exclusion criteria | 8

BASELINE CHARACTERISTICS:
Population: 23 Females participated
Arm/Group | Interventional/Observational
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years]
  Age | 27.4 [20 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23
Skin color according to Fitzpatrick Scales [Count of Participants; unit: Participants] — The Fitzpatrick Scale is a subjective description and categorization of skin color. The categories range from Type I (Light, Pale White) to Type VI (Black, Very Dark, Brown to Black). The scale was originally designed to describe the risk of sunburn. The Fitzpatrick Scale is similar to the Monk Scale. Both are subjective scales of skin color and are used when assessing the potential transdermal effect of melanin.
  Participants
    Type I Skin Color | 2
    Type II Skin Color | 6
    Type III Skin Color | 12
    Type IV Skin Color | 2
    Type V Skin Color | 0
    Type VI Skin Color | 1

OUTCOME MEASURES:

1. Primary Outcome: Fetal Oxygen Levels
Description: Assessment of the adequacy of fetal signals from both internal and external fetal oxygen sensors.
Time Frame: During labor
Population: All 23 subject files were analyzed. Of the 23 participants who completed the monitoring period, 15 were considered to have adequate paired data for analysis of fetal signal.
Measure: Count of Participants; unit: Participants
Groups:
- Interventional/Observational: The internal and external oxygen sensors will be used to record fetal oxygen during active labor. Dual fetal oxygen sensors were used: Placement of both internal and external fetal oxygen sensors to record fetal signals.
Arm/Group | Interventional/Observational
Number analyzed (Participants) | 23
Participants | 15

2. Primary Outcome: Adverse Events
Description: Rate of device-related adverse events such as erythema or rash on the maternal abdomen at the location of the sensor. Note: In this study, use of the device provides additional clinical information, but clinical judgement is based on standard fetal monitoring, including cardiotocography, and investigators are blinded to oximetry readings. The maternal skin at the sensor site will be examined intra and postpartum.
  Rate of device-related adverse events such as erythema or rash on the maternal abdomen at the location of the sensor.
Time Frame: During labor
Measure: Number; unit: participants
Arm/Group | Interventional/Observational
Number analyzed (Participants) | 23
participants | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during the day of participation. Participation was not to exceed 6 hours.
Description: This study was deemed non-significant risk because Investigators were blinded to the fetal oxygen levels; therefore, no sensor data (internal or external) would be used to change clinical decision-making. There were no adverse events or serious adverse events in this study.
Arm/Group | Interventional/Observational
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
This was a research and development study designed to determine if the Lumerah system needed additional modifications to enhance the fetal signal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05147584/Prot_SAP_001.pdf